CLINICAL TRIAL: NCT00070577
Title: Influence of Age and Sex on Alcohol Metabolism and Acute Responses
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030283; 03-AA-0283
Record Dates: First submitted 2003-10-03; First posted 2003-10-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-05-03

CONDITIONS: Metabolism
Keywords: Alcohol Clamp; Pharmacokinetics; Pharmacodynamics; Alcohol; Metabolism; Response; Age; Sex; Healthy Volunteer; HV
MeSH Terms: conditions — Coitus

SUMMARY:
This study will examine age and sex differences in alcohol metabolism and the effects of alcohol. Men and women differ in their ability to metabolize alcohol, possibly due to differences between men and women in lean body mass, liver size, or the activity of enzymes that act on alcohol in the liver. Also, older men and women are thought to be more sensitive to alcohol, although the reasons for this are not clear.

Healthy men and women between 21 and 25 years of age and between 55 and 65 years of age who are social drinkers may be eligible for this study. Candidates will be screened with questionnaires about their general and mental health, alcohol use, and family history of alcohol use and problems. They will have a physical examination, electrocardiogram (EKG), routine blood tests, urinalysis to test for drugs of abuse, and a blood test to study the gene responsible for enzymes that metabolize alcohol. Younger women will have a urine pregnancy test and older women will have a test to confirm post-menopausal status.

Participants will have two study sessions at the NIH Clinical Center outpatient clinic. They come to the clinic by taxi and, upon arrival, take a breathalyzer test for any measurable alcohol levels. They are then given breakfast, after which two catheters (plastic tubes) are placed, one in a vein in each arm. One tube is used to collect blood samples for measuring hormone levels; the other is for infusing alcohol. The infusion is adjusted so that the breath alcohol level is held constant for about 3 hours at a moderate level. Baseline measurements are taken before the infusion begins. During and after the infusion, the participants fill out questionnaires about their moods and feelings. Breath alcohol level and heart rate measurements are monitored frequently. After the test, participants remain in the clinic until their breath alcohol level drops below 0.02 g/L (generally 2 to 3 hours after the infusion stops). They are given lunch and then sent home in a taxi.

Participants also undergo a dual energy x-ray absorptiometry (DEXA) scan to determine lean body mass and a magnetic resonance imaging (MRI) scan of the abdomen to determine liver size. For the DEXA scan, the subject lies still on a table for about 30 minutes while the whole body is scanned using a small amount of radiation. For the MRI, the subject lies in a narrow metal cylinder (the scanner) about 30 minutes for the scan.

DETAILED DESCRIPTION:
Previous studies, including our studies using the alcohol clamp, have shown that alcohol pharmacokinetics differ between women and men. Some of the factors that may contribute to these sex differences in absorption, distribution and metabolism include variation in lean body mass (and total body water), liver size and differences in activity or capacity of alcohol metabolizing enzymes in the stomach and livers of women and men. A fundamental difference between men and women is in the levels of the sex hormones estrogen and testosterone, which can influence several of the above factors. Sex differences in alcohol pharmacokinetics, and estrogen itself, have been postulated as determinants of the increased susceptibility of women to alcohol-related liver disease. An additional area of interest is sex- and age-related differences in sensitivity to the effects of alcohol. The elderly are thought to be more sensitive to alcohol and show greater impairment than younger individuals. However, it is not clear if these changes are due to pharmacokinetic or pharmacodynamic factors.

The objectives of this project are (I) to evaluate the influence of age and sex on alcohol elimination rates in men and women, and (II) to determine the influence of age and sex on the initial response and acute adaptation to alcohol on measures of subjective perceptions of alcohol effects and heart rate. This study will be conducted in 24 young and 24 older participants, with equal numbers of males and females in each group. Comparison of alcohol elimination rates across these groups and correlation with liver volume and sex steroid levels will provide a means to examine the influence of sex hormones, estrogen and testosterone, in age-related and sex-related differences in alcohol metabolism and liver volume. This study will examine age- and sex- related differences in response to alcohol on subjective measures of intoxication and mood, as well as on heart-rate and psychophysiological responses to emotional visual stimuli (pictures). This study will also evaluate the effect of acute alcohol administration on gene expression in peripheral blood cells. Findings from these studies will provide important new data regarding the role of sex steroids (estrogen and testosterone) on the metabolism of alcohol, and a better understanding of age- and sex-related differences in metabolic processes that may underlie medically important differences in the responses of individuals to alcohol.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will be conducted in social drinkers with no current or past history of alcohol dependence or alcohol abuse. Inclusion criteria include:

1. Male and female participants between 21-25 years or 55-65 years of age.
2. Good health as determined by medical history, physical exam, EKG and lab tests.
3. Current non-smokers. Participants who quit smoking for over 1 year can be included.
4. Family-history negative, i.e., no family history of alcoholism in the first-or second-degree.
5. Young women will have normal menstrual cycles and will be tested during the follicular phase of their cycle (within 7 days of offset of menses) and must have a negative urine pregnancy (hCG) test at the start of each study session.
6. Older women will be post-menopausal, with cessation of menses for at least 12 months prior to enrollment into the study, and a serum follicle stimulating hormone (FSH) level greater than 40 IU/L.
7. All participants must report the absence of flushing either currently or in the past, based on the Alcohol Flushing Questionnaire, assessed during screening.
8. Participants must have no ferromagnetic objects in their bodies which might be adversely affected by MRI (e.g. surgical clips; metal fragments in any part of the body; cardiac or neurological pacemaker; cochlear or eye implant) - any doubt about presence of these objects will result in exclusion from this study.

EXCLUSION CRITERIA:

1. Current or prior history of any disease, including cardiovascular, respiratory, gastrointestinal, hepatic, renal, endocrine, or reproductive disorders, or a positive hepatitis or HIV test at screening.
2. Current history of Axis-I psychiatric illness.
3. Current or prior history of any alcohol or drug dependence or abuse, as well as non-drinkers (alcohol-naive individuals or current abstainers).
4. Alcohol use exceeding 14 drinks/week for males and 7 drinks/week for females, and use of more than 4 drinks on any one occasion in the 6 months prior to the study.
5. Positive result on urine drug screen.
6. Pregnancy or intention to become pregnant for women. Female participants will undergo a urine beta-hCG test to ensure they are not pregnant.
7. Use of oral contraceptive pills in younger female participants and use of hormone replacement therapy in older female participants.
8. Menstrual cycle irregularities in younger female participants.
9. Use of prescription or OTC medications known to interact with alcohol within 2 weeks of the study. These include, but may not be limited to: isosorbide, nitroglycerine, benzodiazepines, warfarin, cough-and-cold preparations which contain anti-histamines, codeine and/or acetaminophen, anti-depressants such as amitriptyline, clomipramine and nefazodone, anti-diabetes medications such as glyburide, metformin and tolbutamide, H2-antagonists for heartburn such as cimetidine and ranitidine, muscle relaxants, pain medicines and anti-inflammatories such as aspirin, ibuprofen, acetaminophen, celecoxib and naproxen, anti-epileptics including phenytoin and phenobarbital and narcotics including darvocet, percocet and hydrocodone. Drugs known to inhibit or induce enzymes that metabolize alcohol should not be used for 4 weeks prior to the study. These include acetaminophen, chlorzoxazone, isoniazid, metronidazole and disulfiram.
10. Exclusions also include herbal preparations containing soy isoflavones (which may have estrogenic properties).
11. Inability to undergo the MRI scan for liver volume due to claustrophobia or anxiety when confined to small spaces such as the magnet bore, or due to the presence of metallic implants.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-09-29; Study Completion 2011-05-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aasmoe L, Aarbakke J. Sex-dependent induction of alcohol dehydrogenase activity in rats. Biochem Pharmacol. 1999 May 1;57(9):1067-72. doi: 10.1016/s0006-2952(99)00003-9. PMID 10796077
- [Background] Ammon E, Schafer C, Hofmann U, Klotz U. Disposition and first-pass metabolism of ethanol in humans: is it gastric or hepatic and does it depend on gender? Clin Pharmacol Ther. 1996 May;59(5):503-13. doi: 10.1016/S0009-9236(96)90178-2. PMID 8646821
- [Background] Ayabe T, Tsutsumi O, Sakai H, Yoshikawa H, Yano T, Kurimoto F, Taketani Y. Increased circulating levels of insulin-like growth factor-I and decreased circulating levels of insulin-like growth factor binding protein-1 in postmenopausal women with endometrial cancer. Endocr J. 1997 Jun;44(3):419-24. doi: 10.1507/endocrj.44.419. PMID 9279518